CLINICAL TRIAL: NCT00303381
Title: A Multicentre, Randomised, Double-blind, Placebo-controlled, Dose-finding Phase II Study of Subcutaneously Administered IFN-beta-1a in the Treatment of Patients With Moderately Active Ulcerative Colitis
Brief Title: Safety and Efficacy of Interferon-Beta-1a (Rebif®) for Treating Subjects With Acute Symptoms of Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono (Industry)
Collaborators: Merck Serono International SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22648
Record Dates: First submitted 2006-03-14; First posted 2006-03-16 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Interferon beta-1a

ARMS (3):
- Interferon-beta-1a, 44 microgram (Experimental)
  Interventions: Drug: Interferon-beta-1a, 44 microgram
- Interferon-beta-1a, 66 microgram (Experimental)
  Interventions: Drug: Interferon-beta-1a, 66 microgram
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon-beta-1a, 44 microgram — Interferon-beta-1a will be administered subcutaneously at a dose of 44 mcg, three times a week up to Week 8.
  Other Names: Rebif®
  Arms: Interferon-beta-1a, 44 microgram
Drug: Placebo — Matching Placebo will be administered subcutaneously, three times a week up to Week 8.
  Arms: Placebo
Drug: Interferon-beta-1a, 66 microgram — Interferon-beta-1a will be administered subcutaneously at a dose of 66 mcg, three times a week up to Week 8.
  Other Names: Rebif®
  Arms: Interferon-beta-1a, 66 microgram

SUMMARY:
The purpose of this study is to determine the safety and efficacy of interferon-beta-1a in subjects with active ulcerative colitis (UC).

ELIGIBILITY:
Inclusion Criteria:

* Moderately active UC, defined as:

  * Diagnosis of UC documented by clinical, radiological and endoscopic or histological findings
  * Proctosigmoidoscopic diagnosis: at least left-sided disease; the extent of the colonic inflammation is to be more than 20 centimeter from the anal verge
  * A flare in disease activity considered moderate in according to the UCSS during the 14 days before initiation of study medication. Moderate disease is defined as a UCSS between 6 and 10 with a UCSS Physician's Global Assessment less than (<) 3 and a proctosigmoidoscopy score of 2 or 3
* At least one previous flare-up of UC
* Maintenance treatment with 5-aminosalicylic acid (5-ASA) at a stable dose for the management of UC is allowed, but not required. The daily dose of 5-ASA has to be stable for at least 4 weeks before Study Day 1 and has to be no more than 3.6 gram/day. This dose has to be maintained throughout the study. Corticosteroids will not be allowed during the study, with the exceptions of inhaled steroids and topical dermatological steroids
* Age ≥18 years, of either sex
* Adequate bone marrow reserve: white blood cells (WBC) greater than (>) 3.5*10^9 per liter (/L), neutrophils >1.5*10 ^9 /L, thrombocytes >100 *10^9 /L, hemoglobin >8.5 gram per deciliter (g/dL)
* Female subjects are to be neither pregnant nor breast-feeding and has to lack childbearing potential, as will be defined by either being post-menopausal or surgically sterile or using a hormonal contraceptive, intra-uterine device, diaphragm with spermicide or not pregnant which will be established by a negative serum or urinary Human chorionic gonadotrophin (hCG) test within 7 days before Study Day 1. A pregnancy test is not required if the subject was post-menopausal or surgically sterile
* Willingness and ability to comply with the protocol for the duration of the study
* Written informed consent, obtained before any study-related procedure not part of the subject's normal medical care, with the understanding that the subject can withdraw consent at any time without prejudice to his or her future medical care

Exclusion Criteria:

* Previous systemic treatment with interferons, immunosuppressive therapy (for example [e.g.], cyclosporin, azathioprine, 6-mercaptopurine) or other biological treatment (e.g. anti- Cluster of differentiation [CD] 4, anti-CD5, anti- Tumour necrosis factor [TNF]-alpha, Interleukin [IL]-10) in the 3 months before Study Day 1
* Any other investigational drug or any experimental procedure in the 4 weeks before Study Day 1
* More than three doses of rectally administered 5-ASA derivatives in the 2 weeks before Study Day 1
* More than two doses of systemically or rectally administered corticosteroids in the 14 days before Study Day 1
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) or antibiotic therapy (e.g. metronidazole) in the 2 weeks before Study Day 1
* Use of codeine, other narcotics, loperamide or opiates after the Screening visit or during the study
* Stool examination positive for enteric pathogens, pathogenic ova, parasites, or Clostridium toxin at Screening
* Need for emergency surgery (uncontrollable hemorrhage, persistent non-inflammatory intestinal obstruction - at the Investigator's discretion - or perforation), elective surgery during the study, or surgery in the 4 weeks before study entry
* Inadequate liver function, defined by a total bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase level >2 times the upper limit of the normal range
* Inadequate renal function, defined by serum creatinine >2.0 milligram per deciliter (mg/dL)
* Histopathological findings of high-grade dysplasia or history of cancer (except carcinoma in situ of the cervix or adequately treated basal cell or squamous cell carcinoma of the skin)
* Known allergies to paracetamol or to any of the ingredients of the medicinal product (that is, the active substance, human serum albumin or mannitol)
* Severe depressive disorder or suicidal ideation, or epilepsy with a history of seizures not adequately controlled by treatment
* Known alcohol or drug abuse within the past 5 years
* Other serious concurrent systemic disorders incompatible with the study (at the Investigator's discretion)
* Severe active infection (at the Investigator's discretion)
* Dependence on a liquid diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2001-12; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with endoscopically confirmed remission | Baseline up to Week 12 or early withdrawal or treatment failure

SECONDARY OUTCOMES:
Percentage of subjects with clinical remission | Baseline up to Week 12 or early withdrawal or treatment failure
Percentage of subjects with clinical remission at Week 8 and 12 | Week 8 and 12
Time to first occurrence of clinical remission | Baseline up to Week 12 or early withdrawal or treatment failure
Time to first occurrence of endoscopically confirmed remission | Baseline up to Week 12 or early withdrawal or treatment failure
Percentage of subjects with clinical remission two weeks after endoscopically confirmed remission | Baseline up to Week 12 or early withdrawal or treatment failure
Percentage of subjects with clinical response | Baseline up to Week 12 or early withdrawal or treatment failure
Time to first occurrence of clinical response | Baseline up to Week 12 or early withdrawal or treatment failure
Change from Baseline in Ulcerative Colitis Scoring System (UCSS) total score and sub-scores at Week 2, 4, 6, 8 and 12 | Baseline, Week 2, 4, 6, 8 and 12
Change from Baseline in Inflammatory Bowel Disease Questionnaire (IBDQ) total score and sub-scores at Week 4, 8 and 12 | Baseline, Week 4, 8 and 12
Percentage of subjects with an increase in IBDQ score of at least 15 points | Baseline up to Week 12 or early withdrawal or treatment failure
Change from Baseline in C-reactive protein level at Week 2, 4, 8 and 12 | Baseline, Week 2, 4, 8 and 12
Changes from Baseline in erythrocyte sedimentation rate at Week 2, 4, 8 and 12 | Baseline, Week 2, 4, 8 and 12
Percentage of subjects with treatment failure | Baseline up to Week 12 or early withdrawal or treatment failure

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Pena Rossi, M.D., Study Director — Merck Serono International SA
Locations (7):
- Research Site, Munich, Germany
- Research Site, Ness Ziona, Israel
- Research Site, The Hague, Netherlands
- Research Site, Singapore, Singapore
- Research Site, Solna, Sweden
- Research Site, Zug, Switzerland
- Research Site, Feltham, United Kingdom

REFERENCES:
- [Result] Pena-Rossi C, Schreiber S, Golubovic G, Mertz-Nielsen A, Panes J, Rachmilewitz D, Shieh MJ, Simanenkov VI, Stanton D, Graffner H. Clinical trial: a multicentre, randomized, double-blind, placebo-controlled, dose-finding, phase II study of subcutaneous interferon-beta-la in moderately active ulcerative colitis. Aliment Pharmacol Ther. 2008 Sep 15;28(6):758-67. doi: 10.1111/j.1365-2036.2008.03778.x. PMID 19145731
- See also: Full FDA approved prescribing information can be found here — http://www.mslifelines.com